CLINICAL TRIAL: NCT05745038
Title: A Single Arm Pilot Trial of a Social Network Intervention (SONATA) for Older Patients With Cancer
Brief Title: A Single Arm Pilot Trial of a Social Network Intervention
Acronym: SONATA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Kah Poh Loh, Associate Professor - Department of Medicine, Hematology/Oncology (SMD), University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UOCPC22065
Record Dates: First submitted 2023-02-15; First posted 2023-02-27 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Cancer
Keywords: geriatric oncology
MeSH Terms: conditions — Neoplasms | interventions — zaleplon

STUDY DESIGN:
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 - SONATA Intervention (Experimental)
  Interventions: Behavioral: SONATA

INTERVENTIONS:
Behavioral: SONATA — The SONATA intervention is composed of five components, network diagnostics, network engagement, opportunity creation, skill building and goal-setting, and feedback, that will be audio-recorded and held over six scheduled sessions.

SUMMARY:
The purpose of this study is to see if a social network support program (SOcial Networks to Activate Trust & Adherence or SONATA) is helpful for older individuals receiving cancer treatment. The SONATA program will last for about 4 months. There are a total of 6 coaching sessions. The first 5 sessions will be held approximately every 1 to 2 weeks. Session 6 or the final session will be held approximately 1 to 2 months after session 5. Each session will last for about 1 to 2 hours.

DETAILED DESCRIPTION:
The objective of this study is to conduct a single arm pilot study to assess the feasibility and acceptability of the SONATA intervention among older patients with advanced cancer. We hypothesize that the SONATA intervention will be feasible [≥70% enrolled patient subjects (excluding those who die during the study) will complete at least 3 of the SONATA sessions] and acceptable [average patient subject general acceptability score ≥4 (range one to five) using the Theoretical Framework of Acceptability questionnaire.]

ELIGIBILITY:
Patient

Inclusion Criteria:

1. Age ≥60 years
2. A diagnosis of advanced or likely incurable cancer, as determined by the primary oncologist
3. Able to speak English
4. Able to provide informed consent

Exclusion Criteria:

1) Any psychiatric or cognitive impairments interfering with participation as determined by the primary oncology team

Network Members:

Inclusion Criteria:

1. Age ≥18 years
2. Identified as a network member by patient subjects (up to 10 network members)
3. Able to speak English
4. Able to provide informed consent.

Exclusion Criteria:

None

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2023-11-29 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility - SONATA Intervention | 20 Weeks
  Number of patients approached who consent
Acceptability- SONATA Intervention | 20 Weeks
  Average general acceptability score using the Theoretical Framework of Acceptability questionnaire. An eight item (range 1 to 5 for each item) psychometrically validated and theoretically informed tool which assesses the following constructs - affective attitude, burden, ethicality, perceived effectiveness, intervention coherence, self-efficacy, opportunity costs, and general acceptability.

SECONDARY OUTCOMES:
Estimate - Social Support | 20 Weeks
  Assessed using the Medical Outcomes Study Social Support Survey. The Medical Outcomes Study Social Support Survey is a 19-item survey (range 1-5 for each item) to assess four domains of emotional/informational support, instrumental support, positive social interaction, and affection; higher scores indicate greater social support. Subjects will be asked about their perceptions of their own social support.
Estimate - Trust in Healthcare Professionals | 20 Weeks
  Assessed using the the Human Connection (THC) Scale. The THC scale is A 16-item scale (range 1 to 4 for each item); higher scores indicate greater trust.
Estimate - Adherence to oral anticancer treatments | 20 Weeks
  Assessed using the Domains of Subjective Extent of Nonadherence (DOSE-Nonadherence). The DOSE-Nonadherence scale is a three-item scale (range from none of the time to every time for each item) with eighteen additional items that assesses reasons for non-adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Kah Poh Loh, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and dataset will be shared upon request from the PI
Supporting Information: Study Protocol
Time Frame: The data will be available for 7 years from accrual of the first subject.